CLINICAL TRIAL: NCT07192029
Title: Balloon Guide Catheter to Optimize Outcomes in Stroke Thrombectomy of the Internal Carotid Artery: a Randomized Controlled Trial
Brief Title: Balloon Guide Catheter to Optimize Outcomes in Stroke Thrombectomy of the Internal Carotid Artery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Fujian Medical University Union Hospital (Other); Zhangzhou Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IAT-BOOST
Record Dates: First submitted 2025-09-08; First posted 2025-09-25 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Stroke
Keywords: Balloon Guide Catheter; Thrombectomy; Internal Carotid Artery
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The experimental group (Experimental)
  Interventions: Procedure: Balloon guide catheter combined with conventional thrombectomy treatment
- The control group (Sham Comparator)
  Interventions: Procedure: Standard guide catheter or neurovascular sheath combined with conventional thrombectomy treatment

INTERVENTIONS:
Procedure: Balloon guide catheter combined with conventional thrombectomy treatment — The experimental group will use balloon guide catheter combined with conventional thrombectomy treatment.
  Arms: The experimental group
Procedure: Standard guide catheter or neurovascular sheath combined with conventional thrombectomy treatment — use standard guide catheter or neurovascular sheath combined with conventional thrombectomy treatment
  Arms: The control group

SUMMARY:
To investigate whether using balloon guide catheter with flow arrest during mechanical thrombectomy, compared to non-flow arrest, improves the rate of first pass expanded Thrombolysis in Cerebral Infarction score (eTICI 2c-3) reperfusion for acute ischemic stroke due to internal carotid artery occlusion

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years;
2. Clinical diagnosis of acute ischemic stroke with internal carotid artery occlusion confirmed by imaging (CTA/MRA/DSA), including isolated intracranial internal carotid artery (I-type), internal carotid artery intracranial segment involving middle cerebral artery (L-type), or internal carotid artery intracranial segment involving middle and anterior cerebral arteries (T-type) (including tandem embolic occlusions of the internal carotid artery C1 or common carotid artery);
3. Baseline NIHSS≥6, and meeting local guidelines for mechanical thrombectomy;
4. Time from onset or last known normal to randomization within 24 hours and proceeding to mechanical thrombectomy;
5. Signed informed consent (or by legal representative).

Exclusion Criteria:

1. Pre-stroke mRS score >2
2. Intracranial hemorrhage shown on imaging;
3. Known or suspected internal carotid artery occlusion caused by dissection or atherosclerosis;
4. Vascular tortuosity preventing the use of balloon guide catheter;
5. Prior stent implantation in the target vessel that would impede the use or removal of mechanical thrombectomy devices;
6. Any other circumstances impeding mechanical thrombectomy implementation;
7. Acute occlusion of multiple vascular territories in bilateral anterior circulation or in both the anterior and posterior circulations confirmed by CTA/MRA;
8. Pregnant subjects;
9. Subjects allergic to contrast agents;
10. Subjects refusing to cooperate or unable to tolerate interventional procedures;
11. Subjects whose expected lifetime are less than 90 days;
12. Midline shift or herniation with ventricular mass effect;
13. Subjects deemed unable to participate in follow-up by investigators;
14. Other situations deemed unsuitable for balloon guide catheter use by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Estimated)
Dates: Start 2025-10-12 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of first-pass reperfusion defined as eTICI 2c-3 reperfusion | Perioperative

SECONDARY OUTCOMES:
Good outcome proportion, defined as mRS score 0-2 | 90 days (±7 days) post-procedure
Ordinal Distribution of mRS Scores (mRS Shift analysis) | 90 days (±7 days)
Change in stroke severity (NIHSS score) | 7 days or discharge (whichever occurs first);
Technical success rate | Perioperative
  Defined as the successful delivery of the guiding catheter to the target vessel and completion of the thrombectomy process without replacing the guiding catheter
Final angiographic reperfusion results (eTICI ≥2b, eTICI ≥2c, eTICI 3) | Perioperative
Reperfusion results (eTICI ≥2b, eTICI 3) | Perioperative
Time from groin puncture to successful reperfusion (eTICI ≥2b, eTICI ≥2c); | Perioperative
Number of mechanical thrombectomy attempts | Perioperative
EQ-5D-5L score | 90 ± 7 days after surgery
Proportion of participants with a Barthel Index score of ≥95 | 90 ± 7 days after surgery

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Zhangzhou Municipal Hospital, Zhangzhou, Fujian
  - Xuanwu Hospital, Capital Medical University., Beijing

IPD SHARING:
Plan to Share IPD: No